CLINICAL TRIAL: NCT02874950
Title: Effect of Exercise Training and Ergonomic Modification on Musculoskeletal Disorders Among Office Workers
Brief Title: Effective Methods of Reducing Lower Back, Neck and Shoulder Pain Among Office Workers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Ardalan Shariat, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPM/TNCPI/1.4.18.1(JKEUPM)/F2
Record Dates: First submitted 2016-08-11; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Musculoskeletal Pain; Low Back Pain
Keywords: Exercise
MeSH Terms: conditions — Musculoskeletal Pain; Low Back Pain; Motor Activity | interventions — Exercise; Ergonomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Office exercise training (Experimental): A package of exercise raining was defined by the researcher and one of the intervention group did it for 6 months.
  Interventions: Other: office exercise training
- Ergonomic modification (Experimental): The ergonomic group, followed 6 months ergonomic modification.
  Interventions: Other: ergonomic modification
- Exercise and ergonomic (Experimental): The mixture group, did 6 months exercise training and also followed 6 months ergonomic modification.
  Interventions: Other: Exercise and ergonomic
- Control (Experimental): Control group did not do any exercise and did not follow any ergonomic modification.
  Interventions: Other: Control

INTERVENTIONS:
Other: office exercise training — The exercise group, did 6 months office exercise training.
  Arms: Office exercise training
Other: ergonomic modification — The ergonomic modification group, followed 6 months modified office ergonomic modification.
  Arms: Ergonomic modification
Other: Exercise and ergonomic — The mixture group, did 6 months exercise training and also followed 6 months modified office ergonomic modification.
  Arms: Exercise and ergonomic
Other: Control — Control group did not do any exercise and did not follow any ergonomic modification.
  Arms: Control

SUMMARY:
Background:Musculoskeletal discomforts (MSD), especially in the neck, lower back and shoulder areas, are some of the most common issues among office workers. The Social Security Organization (SOCSO) in Malaysia caps number of cases involving musculoskeletal injuries at a maximum of 10,000 per year.

Objectives: The primary aims of this research were to: 1. Measure the prevalence of MSD in a sample of office workers; 2. Test effective methods of reducing lower back, neck and shoulder pain in this sample by training exercise, or ergonomics modification, or both of them; and 3. Assess discomfort scores and the range of motion of the lower back, neck and shoulder muscles among the office workers after undertaking the different methods for a period of 6 months.

Methods: In a true experimental design, from 10,000 staff in Telecom Malaysia,onehundred and forty two office workers (of whom 50 were male), aged 20-50 y, were allocated randomly, from 3 different locations (Bangsar, Puchung, and Damansara), to one of three intervention groups (receiving training exercise, receiving modified ergonomics, receiving a combination of exercise and ergonomics modification) and a control group (receiving none of these interventions). The Cornell MSD Questionnaire was used to measure musculoskeletal discomforts, with focus on pain severity, before treatment and after 2, 4 and 6 months of the interventions. The range of motion (ROM) of the hip, neck, shoulder and knee were measured by a 12 inch goniometer, and the Borg CR10 scale was used to measure the perceived exertion of training exercises. The rapid office strain assessment (ROSA) questionnaire was used to assess the strain associated with office work. Height and weight were also measured to calculate the body mass index (BMI).

DETAILED DESCRIPTION:
It is expected that, 6 months intervention including exercise training, ergonomic modification and mixture of these 2 intervention, maybe can decrease the severity of pain in lower back, neck and shoulder among office workers.

ELIGIBILITY:
Inclusion Criteria:

* Working in office

Exclusion Criteria:

* Any physical or mental disease any surgery in background any limitation by Dr

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2016-03; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Measuring the prevalence of musculoskeletal disorder By Cornell questionniare | Baseline
  The Cornell MSD Questionnaire was used to measure musculoskeletal discomforts.

SECONDARY OUTCOMES:
Measure the effects of exercise training on decrease the musculoskeletal disorder by measuring the range of motion in neck, shoulder and lower back, and severity of pain will be measured by Cornell questionniare | Change from Baseline musculoskeletal disorder at 6 months
  range of motion was measured by Goniometer.

IPD SHARING:
Plan to Share IPD: Undecided
We have not decided about it yet.

REFERENCES:
- [Derived] Shariat A, Cleland JA, Danaee M, Kargarfard M, Sangelaji B, Tamrin SBM. Effects of stretching exercise training and ergonomic modifications on musculoskeletal discomforts of office workers: a randomized controlled trial. Braz J Phys Ther. 2018 Mar-Apr;22(2):144-153. doi: 10.1016/j.bjpt.2017.09.003. Epub 2017 Sep 6. PMID 28939263